CLINICAL TRIAL: NCT04373109
Title: Stroke Rehabilitation Outcome During COVID-19 Lockdown
Acronym: SROCL
Status: Completed | Type: Observational
Sponsor: Jeremia Held (Other)
Responsible Party: Sponsor-Investigator, Jeremia Held, Dr., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: BASEC-Nr. 2020-00761
Record Dates: First submitted 2020-04-16; First posted 2020-05-04 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Stroke; Rehabilitation; COVID-19; Cohort Studies
MeSH Terms: conditions — Stroke; COVID-19 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-group study: Assessment of intensity of rehabilitation therapy, daily life upper limb use, physical activi-ty engagement, patient-reported quality of life, and motor outcome after stroke
  Interventions: Behavioral: Observation

INTERVENTIONS:
Behavioral: Observation — Observation of intensity of rehabilitation therapy, daily life upper limb use, physical activi-ty engagement, patient-reported quality of life, and motor outcome after stroke

SUMMARY:
COVID-19 has a big impact on individuals and society as a whole. Especially persons with (multiple) comorbidities such as stroke are affected. The impact of COVID-19 on stroke rehabilitation delivery and stroke patients' functioning is unclear.

DETAILED DESCRIPTION:
With 16'000 patients hospitalized and with new permanent disability in approximately 7'000 individuals every year in Switzerland, stroke has a major impact on quality of life and is an enormous socioeconomic burden. Virtually all patients receive inpatient rehabilitation in the sub-acute phase poststroke. However, also in the later phases poststroke, patients receive rehabilitation interventions in outpatient rehabilitation clinics and private practices, with goal to improve or maintain their functional capacity.

Currently, Switzerland finds itself in an extraordinary situation. The Federal Council has issued a series of measures aimed at the population, organizations and institutions, and the cantons. The aim is to curb the spread of the coronavirus and assure the provision of healthcare. The people are invoked to stay at home and only leave the home if absolutely necessary. If they are over the age of 65 or have an underlying medical condition, the Federal Council strongly recommend that you stay at home under any circumstances unless you have to go to the doctor.

With the recommendation of the Swiss Federal Council almost all stroke patients belong to the group who should stay home. Furthermore, all outpatient rehabilitation clinics have reduced the interventions to a minimum. It is unknown how a sudden stop of rehabilitation influences the stroke patients' functional capacities and their perceived quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or haemorrhagic stroke, confirmed by MRI-DWI and/or CT
* Participating in a stroke research project before the Lockdown (ESTREL - BASEC Nr. 2018-02021/ RE-USE - BASEC-Nr. 2017-01070)
* Age 18 years or older
* Verbal and written informed consent of the patient after participants' information

Exclusion Criteria:

* Severe communication or cognitive deficits, that cause inability to follow the procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Rehabilitation data | 3 month after start lockdown
  Nature of rehabilitation therapy, and number and duration of rehabilitation therapy sessions
Motor Activity Log - 14 Item Version | 3 month after start lockdown
  Patient-reported upper limb use in daily life
International Physical Activity Questionnaire | 3 month after start lockdown
  Patient-reported engagement in physical activity in daily life
Patient-Reported Outcomes Measurement Information System - 29 Version | 3 month after start lockdown
  Patient-self-assessment comprising the following categories: 1) physical function, 2) anxiety, 3) depression, 4) fatigue, 5) sleep disturbance, 6) ability to participate in social roles and activities, 7) pain interference and 8) pain intensity

SECONDARY OUTCOMES:
Global Rating of Perceived Changes (physical activity engagement and upper limb use) | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 3 months after lockdown, 6 months after lockdown
  Patient-reported global rating of physical activity engagement and upper limb use in daily life
Fatigue Severity Scale | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 3 months after lockdown, 6 months after lockdown
  Self-reported questionnaire regarding severity of fatigue and its influence on the performance of daily life activities
Hospital Anxiety and Depression Scale | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 3 months after lockdown, 6 months after lockdown
  Depression and anxiety
Montreal Cognitive Assessment | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 3 months after lockdown, 6 months after lockdown
  Assesses cognitive functions
Functional Ambulation Categories | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 3 months after lockdown, 6 months after lockdown
  Classification regarding the ability to walk independently, with or without a walking aid and takes the type of walking surface into account
Ten-Meter Walk Test | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 3 months after lockdown, 6 months after lockdown
  Gait speed and cadence
Rivermead Mobility Index | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 3 months after lockdown, 6 months after lockdown
  Measures the ability of patients to make postural adjustments (e.g, move in bed), transfer (e.g. be-tween bed to chair), walk, and use stairs
Activities-specific Balance Confidence Scale | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 3 months after lockdown, 6 months after lockdown
  Self-reported measure in which patients rate how confident they are in maintaining balance when performing 16 daily life tasks
Fugl-Meyer Motor Assessment | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 3 months after lockdown, 6 months after lockdown
  Upper and lower limb motor function
Action Research Arm Test | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 3 months after lockdown, 6 months after lockdown
  Upper limb capacity
modified Rankin Scale | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 3 months after lockdown, 6 months after lockdown
  Global disability
National Institutes of Health Stroke Scale | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 3 months after lockdown, 6 months after lockdown
  Neurological impairments
Rehabilitation data | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 6 months after lockdown
  Nature of rehabilitation therapy, and number and duration of rehabilitation therapy sessions
Motor Activity Log - 14 Item Version | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 6 months after lockdown
  Patient-reported upper limb use in daily life
International Physical Activity Questionnaire | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 6 months after lockdown
  Patient-reported engagement in physical activity in daily life
Patient-Reported Outcomes Measurement Information System - 29 Version | 4 weeks after lockdown ("extraordinary situation" as defined by the Swiss law), 6 months after lockdown
  Patient-self-assessment comprising the following categories: 1) physical function, 2) anxiety, 3) depression, 4) fatigue, 5) sleep disturbance, 6) ability to participate in social roles and activities, 7) pain interference and 8) pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Andreas R Luft, Prof, Study Chair — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided